CLINICAL TRIAL: NCT01848145
Title: Rapid Infusion of Ofatumumab in Patients With Previously Treated Chronic Lymphocytic Leukemia, a Phase II Trial
Brief Title: Rapid Infusion of Ofatumumab in Patients With Previously Treated Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: GlaxoSmithKline (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI CLL 18
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Ofatumumab; Rapid Infusion
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ofatumumab (Experimental): Rapid Infusion of Ofatumumab
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — The first dose of ofatumumab administered on Day 1 will be 300 mg to minimize infusion reactions. If the initial 300 mg dose of ofatumumab is well-tolerated, without occurrence of any infusion-associated AEs of >= grade 3, on Day 3 ofatumumab will increase to 1000 mg IV. If the Day 3 dose was well-tolerated (i.e., no infusion-associated AE >= grade 3), on Day 8 the ofatumumab dose will escalate to 2000 mg IV. To achieve the primary endpoint for this study, 20% of the 2000 mg ofatumumab dose only will be administered over the first 30 minutes and if tolerated the remaining 80% of the dose will be infused over the remaining 1.5/hours of each treatment. Ofatumumab doses, weeks 3-8, will remain at 2000 mg IV with no further dose escalations. If the Day 8 (Week 2) dose is tolerated all subsequent doses may be infused in the same manner.
  Other Names: Arzerra

SUMMARY:
This is a Phase II, single-arm study of ofatumumab investigating the safety of an accelerated infusion schedule of ofatumumab in patients who have received at least one prior therapy for CLL. The primary endpoint is to evaluate the number of subjects able to complete infusion number 3 (2000 mg) within 15 minutes of the planned time.

DETAILED DESCRIPTION:
The purpose of this study is to develop an accelerated infusion regimen that allows ofatumumab to be delivered in a safe manner while minimizing the time required administering the treatment. We hypothesize there will be fewer infusion-related reactions using the proposed dose-dense approach the first week before accelerating the rate of infusion.

ELIGIBILITY:
Inclusion Criteria:

1. CD20+ B-cell chronic lymphocytic leukemia (B-CLL) according to International Workshop on CLL Working Group (IWCLL WG) Diagnostic Criteria.
2. Have received at least one prior therapy for CLL.

   •If previously treated with ofatumumab must have achieved at least a partial response (PR) and maintained PR for >= 6 months.
3. Requires treatment according to IWCLL-Working Group guidelines.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) <=1.
5. Laboratory parameters <=7 days prior to treatment initiation:

   1. Creatinine <= 1.5 mg/dL upper limit normal (ULN)
   2. Aspartate amino transferase (AST) or alanine amino transferase (ALT) <= 3.0 x ULN
   3. Alkaline phosphatase (ALP) <= 3.0 x ULN
   4. Total Bilirubin level of < 1.5 mg/dL x the institutional ULN unless secondary to Gilbert's disease (or pattern consistent with Gilbert's)
6. Hepatitis B sAg negative and HepB cAb negative. Note: Patients who are HepB sAg negative but are HepB cAb positive (regardless of HepB sAb status) will NOT be allowed.
7. Women of childbearing potential must have a negative serum pregnancy test performed <=72 hours prior to start of treatment. Women of childbearing potential or men with partners of childbearing potential must use effective birth control measures during treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately.
8. Accessible for treatment and follow-up.
9. Able to understand the nature of this study, give written informed consent prior to study entry, and comply with study requirements.
10. No prior antibody therapy for CLL within the previous 3 months.

Exclusion Criteria:

1. Previous treatment with ofatumumab that resulted in a Grade 3 or 4 infusion reaction.
2. Treatment for CLL within last 4 weeks. (Patients who have received steroids or IVIG for autoimmune complications of CLL are eligible).
3. Current active hepatic or biliary disease (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases, or stable chronic liver disease, per assessment by the treating physician).
4. Active bacterial or viral infection or infection requiring intravenous antibiotic treatment at the time of accrual.
5. Central nervous system lymphoma/CLL.
6. Transformation of CLL to aggressive non-Hodgkin lymphoma (NHL) (i.e., Richter's transformation).
7. History of other malignancy <= 2 years of study entry which could affect compliance with the protocol or interpretation of results. History of curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix, low grade, early-stage, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ (DCIS) of the breast treated with curative intent, are generally eligible.
8. Active hepatitis B or C or known HIV positive.
9. Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to visit 1, whichever is longer.
10. History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae.
11. Clinically significant cardiac disease including unstable angina, acute myocardial infarction (within 6 months of enrollment), congestive heart failure (NYHA III-IV), and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities.
12. Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Flinn, MD, PhD, Study Chair — SCRI Development Innovations, LLC
Locations (6):
- United States (6):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Florida Cancer Specialists-South, Fort Myers, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Oncology Hematology Associates, Cincinnati, Ohio
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee

REFERENCES:
- [Derived] Donnellan W, Berdeja JG, Shipley D, Arrowsmith ER, Wright D, Lunin S, Brown R, Essell JH, Flinn IW. A Phase II Trial Evaluating the Safety of Rapid Infusion of Ofatumumab in Patients with Previously Treated Chronic Lymphocytic Leukemia. Oncologist. 2017 Oct;22(10):1156-e111. doi: 10.1634/theoncologist.2017-0236. Epub 2017 Jul 7. PMID 28687625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between July 2013 and June 2015, 34 subjects with at least one prior therapy for Chronic Lymphocytic Leukemia (CLL) were enrolled at 5 investigational sites in the U.S.
Groups:
- Ofatumumab Accelerated Infusion: Ofatumumab administered by intravenous (IV) infusion. .
  * Infusion 1 (Week 1, Day 1): 300 mg IV starting at 3.6 mg/hr and doubling every 30 minutes until reaching a rate of 240 mg/hr. (Planned infusion time: 226 minutes) If tolerated, patients receive Infusion 2.
  * Infusion 2 (Week 1, Day 3): 1000 mg IV starting at 50 mg/hr and doubling every 30 min until reaching a rate of 80 mg/hr. (Planned infusion time: 167 minutes) If tolerated, patients receive Infusion 3.
  * Infusion 3 (Week 2, Day 1): 2000 mg IV, 20% to be given for 30 minutes and, if tolerated, the remaining 80% to be infused over the next 90 minutes. (Planned infusion time: 120 minutes)
  * Weeks 3-8: If 2000mg dose is tolerated, subsequent infusions will be given weekly in the same manner. Assessments will be done at week 12; responding patients can continue receiving the 2000 mg IV infusion monthly for 4 months up to week 28.
Period: Infusion 1: Week 1, Day 1 - 226 Minutes
Arm/Group | Ofatumumab Accelerated Infusion
Started | 34
Completed Within 15min of Infusion Time | 1 (Number of patients who completed within 15 minutes (min) of infusion time.)
Completed | 33 (Includes participants that completed Infusion 1 and proceeded to the next infusion, Infusion 2.)
Not Completed | 1
Not completed — Adverse Event | 1
Period: Infusion 2: Week 1, Day 3 - 167 Minutes
Arm/Group | Ofatumumab Accelerated Infusion
Started | 33
Completed Within 15min of Infusion Time | 24
Completed | 31 (Includes participants that completed Infusion 2 and proceeded to the next infusion, Infusion 3.)
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Disease Progression | 1
Period: Infusion 3: Week 2, Day 1 - 120 Minutes
Arm/Group | Ofatumumab Accelerated Infusion
Started | 31
Completed Within 15min of Infusion Time | 26
Completed (Includes participants that completed Infusion 3 and proceeded to subsequent infusions.) | 30
Not Completed | 1
Not completed — Adverse Event | 1
Period: Subsequent Infusions: Weeks 3-8
Arm/Group | Ofatumumab Accelerated Infusion
Started | 30
Completed | 20
Not Completed | 10
Not completed — Disease Progression | 6
Not completed — Withdrawal by Subject | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Ofatumumab Accelerated Infusion: Ofatumumab administered by intravenous (IV) infusion. The goal is to complete infusion #3 within 120 minutes (+/- 15 minutes).
  * Infusion 1 (Week 1, Day 1): 300 mg IV starting at 3.6 mg/hr and doubling every 30 minutes until reaching a rate of 240 mg/hr. (Planned infusion time: 226 minutes) If tolerated, patients receive Infusion 2.
  * Infusion 2 (Week 1, Day 3): 1000 mg IV starting at 50 mg/hr and doubling every 30 min until reaching a rate of 80 mg/hr. (Planned infusion time: 167 minutes) If tolerated, patients receive Infusion 3.
  * Infusion 3 (Week 2, Day 1): 2000 mg IV, 20% to be given for 30 minutes and, if tolerated, the remaining 80% to be infused over the next 90 minutes. (Planned infusion time: 120 minutes)
  * Weeks 3-8: If 2000mg dose is tolerated, subsequent infusions will be given weekly in the same manner. Assessments will be done at week 12; responding patients can continue receiving the 2000 mg IV infusion monthly for 4 months up to week 28.
Arm/Group | Ofatumumab Accelerated Infusion
Number analyzed (Participants) | 34
Age, Customized [Median (Full Range); unit: years] | 70 [53 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17
Race/Ethnicity, Customized [Number; unit: participants]
  White | 33
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Who Complete an Accelerated Infusion Regimen Within 15 Minutes of the Planned 2-hour Treatment.
Description: Defined as percent of patients who are able to complete the Day 8 (2000 mg IV Ofatumumab) infusion within 15 minutes of the planned 2-hour treatment goal.
Time Frame: At Week 2, Day 1 of therapy
Population: Patients who completed Infusion #3 within the 2 hour treatment goal.
Measure: Number; unit: percentage of participants
Groups:
- Ofatumumab Accelerated Infusion: Ofatumumab administered by intravenous (IV) infusion.
  * Infusion 1 (Week 1, Day 1): 300 mg IV starting at 3.6 mg/hr and doubling every 30 minutes until reaching a rate of 240 mg/hr. (Planned infusion time: 226 minutes) If tolerated, patients receive Infusion 2.
  * Infusion 2 (Week 1, Day 3): 1000 mg IV starting at 50 mg/hr and doubling every 30 min until reaching a rate of 80 mg/hr. (Planned infusion time: 167 minutes) If tolerated, patients receive Infusion 3.
  * Infusion 3 (Week 2, Day 1): 2000 mg IV, 20% to be given for 30 minutes and, if tolerated, the remaining 80% to be infused over the next 90 minutes. (Planned infusion time: 120 minutes)
  * Weeks 3-8: If 2000mg dose is tolerated, subsequent infusions will be given weekly in the same manner. Assessments will be done at week 12; responding patients can continue receiving the 2000 mg IV infusion monthly for 4 months up to week 28.
Arm/Group | Ofatumumab Accelerated Infusion
Number analyzed (Participants) | 31
percentage of participants | 84

2. Secondary Outcome: Duration of Time to Complete Individual Infusions of an Accelerated Infusion Schedule of Ofatumumab
Description: Defined as the actual mean infusion times, in minutes, for patients to complete a schedule of 3 infusions with the goal of completing Infusion #3 within 15 minutes of the planned 2-hour treatment time.
Time Frame: Week 1 - Days 1 and 3, and Week 2, Day 1
Population: Includes all treated participants. 1 participant discontinued treatment after Infusion # 1 but prior to Infusion #2. 2 participants discontinued treatment after Infusion #2 but prior to Infusion #3
Measure: Mean (Full Range); unit: minutes
Arm/Group | Ofatumumab Accelerated Infusion
Number analyzed (Participants) | 34
minutes
  Infusion #1: planned 226 minutes | 316 [156 to 475]
  Infusion #2: planned 167 minutes: number analyzed (Participants) | 33
  Infusion #2: planned 167 minutes | 185 [130 to 285]
  Infusion #3: planned 120 minutes: number analyzed (Participants) | 31
  Infusion #3: planned 120 minutes | 126 [78 to 246]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Defined as the percent of patients having a complete or partial response (CR or PR) assessed by International Workshop on CLL Working Group (IWCLLWG) Diagnostic Criteria (Hallek et al., 2008). CR = (a) Peripheral blood lymphocytes below 4000/µl; (b) Absence of significant lymphadenopathy by physical exam or radiographic scans (c) No hepatomegaly or splenomegaly; (d) Absence of constitutional symptoms; and blood counts above specified values. PR = (a) Decreased blood lymphocytes by 50% or more from the value prior to therapy;(b) No increase in any lymph node, and no new enlarged lymph node. Progressive Disease (PD) = An increase in 50% or more in greatest determined diameter of any previous site. Stable Disease (SD) = No evidence of CR or PR and no evidence of progressive disease.
Time Frame: At weeks 12 and 28
Population: All evaluable patients. 3 patients discontinued prior to assessment.
Measure: Number; unit: percentage of patients
Arm/Group | Ofatumumab Accelerated Infusion
Number analyzed (Participants) | 31
percentage of patients
  ORR | 19
  PR | 19
  SD | 71
  PD | 10

4. Secondary Outcome: Progression Free Survival
Description: Defined as the time from first treatment until objective tumor progression or death from any cause.
Time Frame: For 28 weeks during therapy then every 3 months for 2 years and every 6 months thereafter.
Population: All patients who received at least 1 dose of protocol treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofatumumab Accelerated Infusion
Number analyzed (Participants) | 34
months | 9.25 [7.39 to 11.83]

5. Secondary Outcome: Overall Survival
Description: Defined as the time from first treatment until death from any cause.
Time Frame: For 28 weeks during therapy then every 3 months for 2 years and every 6 months thereafter.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofatumumab Accelerated Infusion
Number analyzed (Participants) | 34
months | NA [29.73 to NA] — At a median follow-up of approximately 24 months overall survival has not been reached.

6. Secondary Outcome: Number of Patients With Infusion-related Reactions Assessed According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v. 4.0.
Description: Patients who received at least 1 dose of protocol treatment either Infusion #1 (300 mg), Infusion #2 (1000 mg) or Infusion #3 (2000 mg) are included in the assessment.
Time Frame: up to 28 weeks
Measure: Number; unit: participants
Arm/Group | Ofatumumab Accelerated Infusion
Number analyzed (Participants) | 34
participants
  Infusion #1: 300 mg | 21
  Infusion #2: 1000 mg | 4
  Infusion #3: 2000 mg | 1

ADVERSE EVENTS:
Time Frame: For 28 weeks during treatment then every 3 months for 2 years, and every 6 months thereafter until disease progression.
Description: All patients who received at least one dose of protocol treatment are included in the safety analysis.
Groups:
- Ofatumumab Accelerated Infusion: Ofatumumab administered by intravenous (IV) infusion. The goal infusion time at Infusion #3 is 120 minutes.
  * Infusion 1 (Week 1, Day 1): 300 mg IV starting at 3.6 mg/hr and doubling every 30 minutes until reaching a rate of 240 mg/hr. (Planned infusion time: 226 minutes) If tolerated, patients receive Infusion 2.
  * Infusion 2 (Week 1, Day 3): 1000 mg IV starting at 50 mg/hr and doubling every 30 min until reaching a rate of 80 mg/hr. (Planned infusion time: 167 minutes) If tolerated, patients receive Infusion 3.
  * Infusion 3 (Week 2, Day 1): 2000 mg IV, 20% to be given for 30 minutes and, if tolerated, the remaining 80% to be infused over the next 90 minutes. (Planned infusion time: 120 minutes)
  * Weeks 3-8: If 2000mg dose is tolerated, subsequent infusions will be given weekly in the same manner. Assessments will be done at week 12; responding patients can continue receiving the 2000 mg IV infusion monthly for 4 months up to week 28.
Arm/Group | Ofatumumab Accelerated Infusion
Serious Adverse Events (participants affected / at risk) | 9/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab Accelerated Infusion (N=34)
Pneumonia (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 2
Bacterial Sepsis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Loss of Consciousness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab Accelerated Infusion (N=34)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 12
Leukopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 7
Anaemia (Blood and lymphatic system disorders) | 9
Lymphopenia (Blood and lymphatic system disorders) | 4
Fatigue (General disorders) | 10
Pyrexia (General disorders) | 7
Chills (General disorders) | 6
Asthenia (General disorders) | 3
Influenza-Like Illness (General disorders) | 2
Oedema (General disorders) | 2
Oedema Peripheral (General disorders) | 2
Nausea (Gastrointestinal disorders) | 8
Abdominal Pain (Gastrointestinal disorders) | 4
Hypoaethesia Oral (Gastrointestinal disorders) | 3
Paraesthesia Oral (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Flushing (Vascular disorders) | 5
Alanine Aminotransferase Increased (Investigations) | 4
Aspartate Aminotransferase Increased (Investigations) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 5
Decreased Appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Insomnia (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 2
Paraesthesia (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Pruritis (Skin and subcutaneous tissue disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Skin Lesion (Skin and subcutaneous tissue disorders) | 2
Urinary Tract Infection (Infections and infestations) | 5
Conjunctivitis (Skin and subcutaneous tissue disorders) | 2
Seasonal Allergy (Immune system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.